CLINICAL TRIAL: NCT06133998
Title: Effects of Incentive Spirometry With and Without Aerobic Exercises on Dyspnea, Exercise Capacity and Quality of Life in Interstitial Lung Disease
Brief Title: Effects of Incentive Spirometry With and Without Aerobic Exercises in Interstitial Lung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0349
Record Dates: First submitted 2023-10-25; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Interstitial Lung Disease
Keywords: shortness of breath ,cough,fatigue.
MeSH Terms: conditions — Lung Diseases, Interstitial; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- incentive spirometry with aerobic exercises (Experimental): Group A: Aerobic exercise (running, jugging, cycling, walking) will be given to the group A for the checking the effect of incentive spirometer
  * In sitting position, for the relaxation of body, patient will take a deep breath.
  * In sitting position, patient will sit on the chair, placed both feet on the floor while bending knee at 90 degree and use the incentive spirometer for the deep breath and check the volume of lung.
  * This schedule will be following supervised exercise training for a minimum 60 minutes 3 days a week in moderate patient,75 minutes in moderate to vigorous patients and 150 minutes in healthy patients
  * We will check the dyspnea of the patient by the borage scale
  * We will check the exercise capacity by the endurance training of respiratory muscles and use the 6 mint walk test
  * We will check the quality of life by the questionnaire.
  Interventions: Device: incentive spirometer with aerobic exercises
- incentive spirometry without aerobic exercises (Active Comparator): Group B: In group B we will check the effects of incentive spirometer without the aerobic exercise.
  * In aerobic exercise following treatment protocol will be involve
  * In sitting position, for the relaxation of body, patient will take a deep breath.
  * In sitting position, patient will sit on the chair, placed both feet on the floor while bending knee at 90 degree and use the incentive spirometer for the deep breath and check the volume of lung.
  * We will check the dyspnea of the patient by the borage scale
  * We will check the exercise capacity by the endurance training of respiratory muscles and use the 6 mint walk test
  * We will check the quality of life by the questionnaire.
  * We will check the chest expansion by measuring tap.
  Interventions: Device: incentive spirometry without aerobic exercises

INTERVENTIONS:
Device: incentive spirometer with aerobic exercises — Group A: Aerobic exercise (running, jugging, cycling, walking) will be given to the group A for the checking the effect of incentive spirometer
  * In sitting position, for the relaxation of body, patient will take a deep breath.
  * In sitting position, patient will sit on the chair, placed both feet on the floor while bending knee at 90 degree and use the incentive spirometer for the deep breath and check the volume of lung. This schedule will be following supervised exercise training for a minimum 60 minutes 3 days a week in moderate patient,75 minutes in moderate to vigorous patients and 150 minutes in healthy patients
  * We will check the dyspnea of the patient by the borage scale
  * We will check the exercise capacity by the endurance training of respiratory muscles and use the 6 mint walk test
  * We will check the quality of life by the questionnaire.
  Arms: incentive spirometry with aerobic exercises
Device: incentive spirometry without aerobic exercises — Group B: In group B we will check the effects of incentive spirometer without the aerobic exercise.
  * In aerobic exercise following treatment protocol will be involve
  * In sitting position, for the relaxation of body, patient will take a deep breath.
  * In sitting position, patient will sit on the chair, placed both feet on the floor while bending knee at 90 degree and use the incentive spirometer for the deep breath and check the volume of lung.
  * We will check the dyspnea of the patient by the borage scale
  * We will check the exercise capacity by the endurance training of respiratory muscles and use the 6 mint walk test
  * We will check the quality of life by the questionnaire.
  * We will check the chest expansion by measuring tap.
  Arms: incentive spirometry without aerobic exercises

SUMMARY:
Effects of Incentive spirometry with and without Aerobic exercises on dyspnea, exercise capacity and quality of life in interstitial lung disease

DETAILED DESCRIPTION:
Interstitial lung disease is the large group of diseases most of which cause progressive scarring of lung tissue. The scarring associated with interstitial lung disease eventually affects participants ability to breathe and get enough oxygen into participants bloodstream. This is occurring by the long term work in dusty places or factories Randomized control trials will be conducted in DHQ hospital Layyah through the convent sampling techniques on patients which will be allocated through convenience sampling technique on 32 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A and group B. After the conventional treatment Group A will be treated with aerobic exercise and Group B will be treated without the aerobic exercise. In group A check the effect of spirometry with aerobic exercise (walking, jogging, running and cycling) and group B check the effect of spirometry without the aerobic exercise and dyspnea by using the 6 mint walk test, Borage scale, PFT, chest expansions and quality of life questionnaire. investigators apply the aerobic exercise by using the spirometer on the interstitial lung diseases patient and check the effectiveness of dyspnea, exercise capacity and quality of life of the patient. Data will be collect by the questioner and Data will be analyzed using SPSS software version 21. After assessing normality of data by Shapiro - wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients18 to 55 years of age (21)
* Both gender(M/F)
* Diagnosed as ILD ( sarcoidosis,acute interstitial pneumonia etc.)on clinical, radiological, and histopathological basis
* All included patients were clinically stable without exacerbations in the past 1 month.

Exclusion Criteria:

* Patients with other significant respiratory disorders such as acute infections, pulmonary tuberculosis, COPD, asthma, bronchiectasis, lung carcinoma, and pneumothorax
* connective tissue disease-associated ILD
* Patients having other co morbid diseases preventing from exercise training, for example, disability due to orthopedic, neurological, and acute cardiac causes
* Physically and mentally unwell to attend the hospital for training
* Already completed or participated in a PR program in the past 1 year

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
FVC (force vital capacity) | 6 weeks
  Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange. Spirometry the most common type of lung function test. It measures how much and how quickly you can move air in and out of your lungs. Measure the values of FVC (force vital capacity) in liters and in predicted % form . Normal value of FVC is 4.75 to 5.5 in male and 3.25 to3.75 in female.
The value of FEV1 | 6 weeks
  Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange. Spirometry the most common type of lung function test. It measures how much and how quickly you can move air in and out of your lungs. Measure the value of FEV1 in liters and in predicted% form. Normal FEV1 in male is3.5to 4.5 and in female is 2.5 to 3.25.
Borg scale | 6 weeks
  This scale use for the measurement of dyspnea (shortness of breath) Borg rating of perceived exertion (RPE) is an outcome measure scale used in knowing exercise intensity prescription. It is used in monitoring progress and mode of exercise in cardiac patients as well as in other patient populations undergoing rehabilitation and endurance training. According to the Borg scale maximum value is 9-10which shows the severe pain level in patient and the moderate pain value is 3-4 the minimum pain is values 1-2 .
6mint walk test | 6 weeks
  This test is performing for the measurement of aerobic capacity and endurance. The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity
Quality of life questioner | 6 weeks
  This questioner is use for measure of physical, psychological and emotional wellbeing life. The QOLQ is a validated and reliable questionnaire that measures an individual's physical, psychological, and social well-being. It consists of a set of questions that cover various aspects of quality of life, such as physical health, emotional well-being, social support, and overall satisfaction with life
chest expansion | 6 weeks
  In this test we use the measuring tape for the measurement of chest mobility. Chest expansion, defined as the difference in thoracic girth after maximum inspiration and maximum expiration, is one indicator of chest wall mobility. As it is measured using a measuring tape, it is a simple, inexpensive, and noninvasive tool for assessing chest mobility.

CONTACTS AND LOCATIONS:
Overall Officials: sumera abdul hameed, Ms, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilyy A, El-Nakhal T, Kadlec J, Bartosik W, Tornout FV, Kouritas V. Preoperative training education with incentive spirometry may reduce postoperative pulmonary complications. Asian Cardiovasc Thorac Ann. 2020 Nov;28(9):592-597. doi: 10.1177/0218492320957158. Epub 2020 Sep 11. PMID 32915659
- [Background] Larson M, Kim MJ. Respiratory muscle training with the incentive spirometer resistive breathing device. Heart Lung. 1984 Jul;13(4):341-5. PMID 6564101
- [Background] Scherer TA, Spengler CM, Owassapian D, Imhof E, Boutellier U. Respiratory muscle endurance training in chronic obstructive pulmonary disease: impact on exercise capacity, dyspnea, and quality of life. Am J Respir Crit Care Med. 2000 Nov;162(5):1709-14. doi: 10.1164/ajrccm.162.5.9912026. PMID 11069801
- [Background] Ho SC, Chiang LL, Cheng HF, Lin HC, Sheng DF, Kuo HP, Lin HC. The effect of incentive spirometry on chest expansion and breathing work in patients with chronic obstructive airway diseases: comparison of two methods. Chang Gung Med J. 2000 Feb;23(2):73-9. PMID 10835801
- [Background] Rondinel TZ, Correa IF, Hoscheidt LM, Bueno MH, Da Silva LM, Reppold CT, Dal Lago P. Incentive spirometry combined with expiratory positive airway pressure improves asthma control and quality of life in asthma: a randomised controlled trial. J Asthma. 2015 Mar;52(2):220-6. doi: 10.3109/02770903.2014.956890. Epub 2014 Sep 2. PMID 25144550